CLINICAL TRIAL: NCT01779908
Title: Role of Vitamin D in the Prevention and Treatment of Diseases Associated With Insulin Resistance
Acronym: VIDIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CHU de Quebec-Universite Laval (Other)
Collaborators: Canadian Diabetes Association (Other); Laval University (Other); Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Claudia Gagnon, MD, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CDA grant no OG-3-12-3681-CG; B12-12-1095
Record Dates: First submitted 2013-01-24; First posted 2013-01-30 (Estimated); Last update posted 2020-07-24 (Actual); Status verified 2020-07

CONDITIONS: Vitamin D-deficient; Insulin-resistant
Keywords: Vitamin D supplementation; Insulin resistance
MeSH Terms: conditions — Insulin Resistance | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D supplementation (Experimental): 5000 IU of vitamin D3 for 6 months
  Interventions: Dietary Supplement: Vitamin D
- Placebo (Placebo Comparator): Placebo pill for 6 months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D
  Arms: Vitamin D supplementation
Other: Placebo
  Arms: Placebo

SUMMARY:
Prospective, randomized and placebo-controlled 6-month trial of vitamin D supplementation in 130 Caucasian and vitamin D-deficient men and women aged 25 years and over. Participants will have abdominal obesity and at least one factor associated with insulin resistance. Participants will be randomized by sex, BMI and age. The primary aim is to compare the effect of daily vitamin D3 (cholecalciferol, 5000 IU) vs. placebo for 6 mo on insulin sensitivity (M-value by the gold standard method, the euglycemic hyperinsulinemic clamp). Secondary aims are to evaluate the effects of vitamin D3 vs. placebo on other indices of glucose metabolism, the lipid profile, blood pressure and anthropometric measurements. Questionnaires on physical activity and sunlight exposure, and a food frequency questionnaire will be administered at 0 and 6 mo to adjust for confounding factors. At 0 and 6 mo, changes in serum 25(OH)D will be correlated with changes in blood markers associated with insulin sensitivity [hs-CRP, inflammatory cytokines (IL-6 and TNF-alpha), adiponectin, leptin, total and undercarboxylated osteocalcin].

This research project intends to test 2 major hypotheses: (1) that vitamin D deficiency plays a causal role in the pathogenesis of insulin resistance in humans; and (2) that vitamin D increases insulin sensitivity.

DETAILED DESCRIPTION:
Part 1: Prospective, randomized and placebo-controlled 6-month trial of vitamin D supplementation in 130 Caucasian and vitamin D-deficient [serum 25(OH)D ≤55 nM] men and women aged 25 years and over with a BMI ≤40 kg/m2. Participants will have abdominal obesity (increased waist circumference of at least 102 cm for men and 88 cm for women) and at least one factor associated with insulin resistance, namely: (1) serum triglyceride levels of at least 1.7 mmol/L or treated dyslipidemia; (2) prediabetes or untreated type 2 diabetes (HbA1c >=5.6% or fasting glucose >=5.6 mmol/L or glucose 2h post OGTT >=7.8 mmol/L); (3) first degree relative with type 2 diabetes; (4) history of gestational diabetes. Participants will be randomized according to sex, BMI (<30 kg/m2 vs. 30 kg/m2 and over) and age (< or >=50 years old). The primary aim is to compare the effect of daily vitamin D3 (cholecalciferol, 5000 IU) vs. placebo for 6 mo on insulin sensitivity (M-value by the gold standard method, the euglycemic hyperinsulinemic clamp). Secondary aims are to evaluate the effects of vitamin D3 vs. placebo on other indices of glucose metabolism (fasting glucose, 2-h plasma glucose post OGTT, HbA1c, insulin sensitivity index (HOMA-IS using fasting glucose and insulin), insulin secretion index (HOMA-B using fasting glucose and C-peptide), insulinogenic index [(C-peptide at 30 min post OGTT - C-peptide at 0 min)/(glucose at 30 min post OGTT - glucose at 0 min)] and disposition index (insulinogenic index x M-value)), the lipid profile, blood pressure and anthropometric measurements (weight, waist and hip circumference, bioimpedance analysis). Questionnaires on physical activity and sunlight exposure, and a food frequency questionnaire will be administered at 0 and 6 mo to adjust for confounding factors. At 0 and 6 mo, biochemical markers associated with insulin sensitivity will be measured (point 2).

Part 2: Mechanistic studies comparing, before and after vitamin D3 supplementation, changes in serum 25(OH)D with changes in blood markers associated with insulin sensitivity [hs-CRP, inflammatory cytokines (IL-6 and TNF-alpha), adiponectin, leptin, total and undercarboxylated osteocalcin].

ELIGIBILITY:
Inclusion Criteria:

* Caucasian men and women
* ≥25 yrs
* vitamin D deficiency [serum 25(OH)D concentration ≤55 nM]
* Abdominal obesity (waist circumference >=102 cm for men and >=88 cm for women) AND at least one factor associated with insulin resistance: (1) fasting serum triglycerides >=1.7 mmol/L or treated dyslipidemia; (2) prediabetes or untreated type 2 diabetes (HbA1c >=5.6% or fasting glucose >=5.6 mmol/L or 2h glucose post OGTT >=7.8 mmol/L); (3) first degree relative with type 2 diabetes; (4) history of gestational diabetes.

Exclusion Criteria:

* Type 2 diabetes under drug therapy
* HbA1c >7%
* BMI >40 kg/m2
* pregnancy or breast-feeding;
* medication influencing vitamin D or glucose metabolism in the last 3 mo
* regular consumption of supplements containing >400 IU/d of vitamin D3 over the last 2 mo;
* renal insufficiency (creatinine clearance <60 ml/min);
* cirrhosis,
* intestinal malabsorption (bypass surgery, celiac disease, etc);
* osteoporosis;
* history of nephrolithiasis;
* hypercalcemia (>2.6 mM);
* hypercalciuria (>0.6 fasting urine Ca/creatinine ratio);
* >5% change in weight in the last 3 mo;
* diseases affecting glucose metabolism (e.g. hyperthyroidism);
* pacemaker (for bioimpedance only);
* inability to provide informed consent and complete questionnaires due to physical or mental problems.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2013-01; Primary Completion 2017-06-02 (Actual); Study Completion 2020-06 (Actual)

PRIMARY OUTCOMES:
Change in peripheral insulin sensitivity assessed by the euglycemic-hyperinsulinemic clamp between placebo and vitamin D groups | 0 and 6 months
  M-value
Change in peripheral insulin sensitivity assessed by the euglycemic-hyperinsulinemic clamp between placebo and vitamin D groups | 0 and 6 months
  M/I ratio

SECONDARY OUTCOMES:
Change in insulin sensitivity indice assessed by fasting- and oral glucose tolerance test between placebo and vitamin D groups | 0 and 6 months
  HOMA2%S
Change in insulin sensitivity indice assessed by fasting- and oral glucose tolerance test between placebo and vitamin D groups | 0 and 6 months
  Matsuda index
Change in insulin secretion indice between placebo and vitamin D groups | 0 and 6 months
  area under the curve for C-peptide
Change in insulin secretion indice between placebo and vitamin D groups | 0 and 6 months
  HOMA2-B
Change in insulin secretion indice between placebo and vitamin D groups | 0 and 6 months
  insulinogenic index
Change in B-cell function between placebo and vitamin D groups | 0 and 6 months
  Disposition index
Change in metabolic markers between placebo and vitamin D groups | 0 and 6 months
  HbA1c
Change in metabolic markers between placebo and vitamin D groups | 0 and 6 months
  Fasting glucose
Change in metabolic markers between placebo and vitamin D groups | 0 and 6 months
  2h glucose post-OGTT
Change in anthropometry between placebo and vitamin D groups | 0 and 6 months
  Weight
Change in anthropometry between placebo and vitamin D groups | 0 and 6 months
  BMI
Change in anthropometry between placebo and vitamin D groups | 0 and 6 months
  waist circumference
Change in anthropometry between placebo and vitamin D groups | 0 and 6 months
  hip circumference
Change in anthropometry between placebo and vitamin D groups | 0 and 6 months
  fat mass by bioimpedance analysis
Change in blood pressure between placebo and vitamin D groups | 0 and 6 months
  Systolic and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Gagnon, Dr., Principal Investigator — CHU de Québec Research Center
Locations (1):
- CHU de Québec, Laval University Research Center, Québec, Quebec, Canada